CLINICAL TRIAL: NCT02250859
Title: An Open-label, Multiple Dose Study to Assess the Pharmacokinetic Profile of Minocycline From FMX-101 Foam (4%) in Male and Female Volunteers
Brief Title: A Pharmacokinetic Study of Minocycline in Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMX101-1
Record Dates: First submitted 2014-09-21; First posted 2014-09-26 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FMX101 Minocycline 4% foam (Experimental): FMX101, 4% applied to the face, upper chest, upper back and shoulders for sixsteen consecutive days in subjects either with acne or with normal skin
  Interventions: Drug: FMX101, Minocycline 4% foam

INTERVENTIONS:
Drug: FMX101, Minocycline 4% foam — FMX101, Minocycline 4% foam to be applied twice daily for 16 consecutive days
  Other Names: FMX101 antibiotic foam

SUMMARY:
The purpose of this study is to assess the pharmakokinetic profile of Minocycline in FMX-101 4% foam product in male and female some of which are with acne

DETAILED DESCRIPTION:
This is an open-label, single-center, non-randomized, multiple-administrations study in males and females, some of which are with acne.

Twelve (12) subjects will be enrolled to receive a daily dose of topical FMX-101 minocycline (4%) foam for sixteen consecutive days.

Each subject will undergo screening procedures within 21 days prior to dosing, to assess his eligibility to participate in the study, including a dermatological assessment of the acne severity and distribution (for subjects with acne).

On Days 1, 2, 3, 7, 9, 11, 14, 16 and 17 blood will be drawn for PK An End-of Study/Safety Follow-up visit will take place on 7-10 days after last dose, which will also include a dermatological assessment of response to treatment

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 35 years (inclusive) of age.
2. Clear skin or facial acne of any severity, currently untreated
3. Otherwise healthy subjects
4. Subjects who provide written informed consent to participate in the study.
5. Women of childbearing potential who are willing to use 2 reliable methods of contraception or practice abstinence during the study period or be surgically sterilized and agree to undergo repeated pregnancy tests.
6. Body Mass Index (BMI) 19.0 to <30.0 kg/m2 and weight ranging between 60-90 kg (males) and 50-85 (females).
7. Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 6 months prior to screening visit
8. Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs, ECG and a physical examination.
9. Shaven facial hair (males)
10. Negative HIV, Hepatitis B and Hepatitis C serology tests at screening.
11. No clinically significant abnormalities in hematology, blood chemistry, or urinalysis lab tests at screening.
12. No known history of alcohol or drug abuse. Negative urinary screen for drugs of abuse determined within 21 days of the start of the study (screening visit).
13. Willingness to minimize exposure to sun for 20 days after first dosing
14. Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study

Exclusion Criteria:

1. Documented history or ongoing symptoms of significant neurological, renal, cardiovascular, respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
2. Known or suspected pregnancy or lactation or planned pregnancy during the study duration (females)
3. Use of topical antibiotics or topical corticosteroids for acne treatment within the past 2 weeks.
4. Use of systemic corticosteroids within the past 4 weeks.
5. Use of systemic retinoids (e.g. isotretinoin) within the past 6 months.
6. Concurrent use of medications known to be photosensitizers because of the possibility of augmented photosensitivity.
7. History or evidence of skin conditions other than acne (eg, eczema) that would interfere with the subject's participation in the study.
8. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol or ibuprofen for symptomatic relief of pain is allowed until 24 hours prior to the study drug administration.
9. Dermatological conditions which might have an effect upon dermal application, e.g.: Psoriasis, mycosis fungoides, widespread acne, facial or back dermatophytosis, severe hyperhydrosis, chronic or recurrent skin infections, ichtyosis
10. Excessive hair in the intended application areas
11. Current or recent (within 1year) drug or alcohol abuse.
12. Known contraindication, hypersensitivity and/or allergy to the study drug or its excipients.
13. Subjects with significant allergic response to other drugs
14. Any acute illness (e.g. acute infection) within 48 hours prior to the first study drug administration, which is considered of significance by the Principal Investigator.
15. Participation in another clinical trial with drugs received within 3 months prior to dosing (calculated from the previous study's last dosing date).
16. Subjects who donated blood in the three months or received blood or plasma derivatives in the six months preceding study drug administration.
17. Subjects unable to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).
18. Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
adverse events | 22-25 days
  AEs will be assessed starting from informed consent signature until end of study)
irritation and local reaction | 16 days
  The application area will be examined for irritation and local reaction
Change from baseline in vital signs | 22-25 days
  sitting BP, HR, RR, oral temperature
Cmax | 16 days
  will be assessed after 1 and 16 days of dosing
Tmax | 16 days
  will be assessed after 1 and 16 days of dosing
AUCT | 16 days
  will be assessed after 1 and 16 days of dosing
T½ | 16 days
  will be assessed after 1 and 16 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Principal Investigator — Sourasky Medical center, Tel-aviv, Israel
Locations (1):
- Sourasky Medical Center, Clinical Research Center, Tel Aviv, Israel